CLINICAL TRIAL: NCT02431260
Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety and Tolerability Study of INCB054329 in Subjects With Advanced Malignancies
Brief Title: An Open-Label, Dose-Escalation Study of INCB054329 in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: As of 31 JAN 2018, the study was terminated by the sponsor due to PK variability.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54329-101
Expanded Access: NCT03896815 (No longer available)
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumors and Hematologic Malignancy
Keywords: solid tumor; lymphoma; BET bromodomain inhibitor; BRD; Diffuse large B-cell lymphoma (DLBCL); Burkitt's lymphoma; c-MYC; colorectal cancer; Non-small cell lung cancer; Pancreatic adenocarcinoma; castration-resistant prostate cancer; breast cancer; NUT midline carcinoma; leukemia; acute myeloid leukemia (AML); myelodysplastic syndrome (MDS); myeloproliferative neoplasms; myelofibrosis (MF); multiple myeloma (MM); MDS/MPN
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Primary Myelofibrosis; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INCB054329 Monotherapy (Experimental)
  Interventions: Drug: INCB054329 Monotherapy

INTERVENTIONS:
Drug: INCB054329 Monotherapy — Initial cohort dose of INCB054329 monotherapy at the protocol-specified starting dose in the treatment group A (TGA), with subsequent cohort escalations in the three treatment groups (TGA, TGB, and TGC) based on protocol-specific criteria

SUMMARY:
This was a study of INCB054329 given to patients with advanced malignancies that were conducted in three treatment groups. Each treatment group had a dose escalation (Part 1) and a dose expansion (Part 3), two of the treatment groups also had an intra-patient dose titration (Part 2).

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of advanced malignancy:

  * Treatment Group A (TGA): Part 1 and Part 2: Any advanced solid tumor or lymphoma; Part 3: Histologically confirmed disease in specific solid tumors and lymphomas
  * Treatment Group B (TGB): Acute Leukemia (Part 3 - acute myeloid leukemia [AML] only), myelodysplastic syndrome (MDS), myelodysplastic /myeloproliferative neoplasms (MDS/MPN) and myelofibrosis (MF)
  * Treatment Group C (TGC): Multiple myeloma
* Progressed following at least 1 line of prior therapy and there is no further approved therapy available that has been demonstrated to prolong survival (including subjects who are intolerant to the approved therapy)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 in Parts 1 and 2 dose escalation and titration, and 0, 1, 2 in Part 3 dose expansion

Key Exclusion Criteria:

* Inadequate hematopoietic, liver, endocrine or renal function
* Receipt of anticancer medications or investigational drugs within the following interval before the first administration of study drug:

  * < 6 weeks for mitomycin-C or nitrosoureas
  * < 5 half-lives or 14 days, whichever is longer, for any investigational agent (for any indication)
  * < 28 days for any antibodies or biological therapies
  * < 5 half-lives for all other anticancer medications, or sponsor approval
* Prior radiotherapy within 2 weeks prior to first dose of study drug
* Untreated brain or central nervous system (CNS) metastases
* Type 1 diabetes or uncontrolled Type 2 diabetes
* Any sign of clinically significant bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Zheng, M.D., Study Director — Incyte Corporation
Locations (12):
- United States (12):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, Medical Center at Mount Zion, San Francisco, California
  - Sarah Cannon Research Institute Research Center, Denver, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Horizon Oncology Center, Lafayette, Indiana
  - John Hopkins, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falchook G, Rosen S, LoRusso P, Watts J, Gupta S, Coombs CC, Talpaz M, Kurzrock R, Mita M, Cassaday R, Harb W, Peguero J, Smith DC, Piha-Paul SA, Szmulewitz R, Noel MS, Yeleswaram S, Liu P, Switzky J, Zhou G, Zheng F, Mehta A. Development of 2 Bromodomain and Extraterminal Inhibitors With Distinct Pharmacokinetic and Pharmacodynamic Profiles for the Treatment of Advanced Malignancies. Clin Cancer Res. 2020 Mar 15;26(6):1247-1257. doi: 10.1158/1078-0432.CCR-18-4071. Epub 2019 Sep 16. PMID 31527168

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 / Treatment Group A: 15 MG QD INCB054329; Part 1 / Treatment Group A: 22.5 MG QD INCB054329; Part 1 / Treatment Group A: 15 MG BID INCB054329; Part 1 / Treatment Group A: 30 MG QD INCB054329; Part 1 / Treatment Group A: 22.5 MG BID INCB054329; Part 1 / Treatment Group A: 20 MG BID INCB054329: Part 1 / treatment group A (TGA): Initial cohort dose of INCB054329 monotherapy at the protocol-specified starting dose in the TGA. Treatment Group A included any advanced solid tumor or lymphoma.
- Part 1 / Treatment Group A: 22.5 MG BID 5/2 INCB054329; Part 1 / Treatment Group A: 25 MG BID 5/2 INCB054329: Part 1 / treatment group A (TGA): Initial cohort dose of INCB054329 monotherapy at the protocol-specified starting dose in the TGA. 5/2=5 days on/2 days off.
  Treatment Group A included any advanced solid tumor or lymphoma.
- Part 1 / Treatment Group A: 22.5 MG BID 4/3 INCB054329: Part 1 / treatment group A (TGA): Initial cohort dose of INCB054329 monotherapy at the protocol-specified starting dose in the TGA. 4/3=4 days on/3 days off. Treatment Group A included any advanced solid tumor or lymphoma.
- Part 1 / Treatment Group A: 22.5 MG BID 7/7 INCB054329; Part 1 / Treatment Group A: 25 MG BID 7/7 INCB054329: Part 1 / treatment group A (TGA): Initial cohort dose of INCB054329 monotherapy at the protocol-specified starting dose in the TGA. 7/7=7 days on/7 days off. Treatment Group A included any advanced solid tumor or lymphoma.
- Part 1 / Treatment Group B: 20 MG BID INCB054329: Part 1 / treatment group B (TGB): Initial cohort dose of INCB054329 monotherapy at the protocol-specified cohort escalation treatment group B (TGB), based on protocol-specific criteria. Treatment Group B included acute leukemia, myelodysplastic syndrome, myelodysplastic/myeloproliferative neoplasms, or myelofibrosis.
- Part 2 / Treatment Group A: 20 MG BID INCB054329: Part 2 / treatment group A (TGA): dose titration was to determine the feasibility of intraparticipant dose titration using Protocol-defined criteria. Treatment Group A included any advanced solid tumor or lymphoma.
- Part 2 / Treatment Group C: 20 mg BID INCB054329: Part 2 / treatment group C (TGC): dose titration was to determine the feasibility of intraparticipant dose titration using Protocol-defined criteria. Treatment Group C included multiple myeloma.
Period: Overall Study
Arm/Group | Part 1 / Treatment Group A: 15 MG QD INCB054329 | Part 1 / Treatment Group A: 22.5 MG QD INCB054329 | Part 1 / Treatment Group A: 15 MG BID INCB054329 | Part 1 / Treatment Group A: 30 MG QD INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 5/2 INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 4/3 INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 7/7 INCB054329 | Part 1 / Treatment Group A: 20 MG BID INCB054329 | Part 1 / Treatment Group A: 25 MG BID 5/2 INCB054329 | Part 1 / Treatment Group A: 25 MG BID 7/7 INCB054329 | Part 1 / Treatment Group B: 20 MG BID INCB054329 | Part 2 / Treatment Group A: 20 MG BID INCB054329 | Part 2 / Treatment Group C: 20 mg BID INCB054329
Started | 4 | 5 | 6 | 5 | 3 | 4 | 4 | 3 | 8 | 8 | 4 | 4 | 10 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 5 | 6 | 5 | 3 | 4 | 4 | 3 | 8 | 8 | 4 | 4 | 10 | 1
Not completed — Subject Decision | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Death | 4 | 4 | 3 | 4 | 2 | 2 | 3 | 1 | 6 | 6 | 3 | 2 | 5 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by the Sponsor | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 4 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Unspecified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants who received at least 1 dose of INCB054329.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 / Treatment Group A: 15 MG QD INCB054329 | Part 1 / Treatment Group A: 22.5 MG QD INCB054329 | Part 1 / Treatment Group A: 15 MG BID INCB054329 | Part 1 / Treatment Group A: 30 MG QD INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 5/2 INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 4/3 INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 7/7 INCB054329 | Part 1 / Treatment Group A: 20 MG BID INCB054329 | Part 1 / Treatment Group A: 25 MG BID 5/2 INCB054329 | Part 1 / Treatment Group A: 25 MG BID 7/7 INCB054329 | Part 1 / Treatment Group B: 20 MG BID INCB054329 | Part 2 / Treatment Group A: 20 MG BID INCB054329 | Part 2 / Treatment Group C: 20 mg BID INCB054329 | Total
Number analyzed (Participants) | 4 | 5 | 6 | 5 | 3 | 4 | 4 | 3 | 8 | 8 | 4 | 4 | 10 | 1 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (4.03) | 54.8 (13.39) | 57.7 (8.50) | 63.6 (7.86) | 68.7 (5.77) | 49.3 (21.73) | 61.5 (12.40) | 68.3 (16.20) | 58.4 (17.55) | 60.9 (14.84) | 50.3 (16.58) | 71.8 (8.77) | 59.3 (14.20) | 66.0 | 60.03 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 3 | 1 | 3 | 2 | 1 | 3 | 4 | 1 | 2 | 7 | 1 | 36
  Male | 2 | 3 | 2 | 2 | 2 | 1 | 2 | 2 | 5 | 4 | 3 | 2 | 3 | 0 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 4 | 5 | 5 | 3 | 3 | 4 | 4 | 3 | 7 | 8 | 4 | 4 | 9 | 1 | 64
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 00 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 5 | 6 | 5 | 3 | 2 | 4 | 3 | 7 | 8 | 4 | 3 | 10 | 1 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 167.3 (8.02) | 172.7 (11.47) | 169.1 (9.80) | 164.6 (10.48) | 172.0 (12.12) | 164.8 (16.52) | 170.8 (16.64) | 174.2 (14.65) | 173.6 (7.05) | 170.5 (12.60) | 179.8 (7.41) | 167.0 (13.29) | 160.8 (10.40) | 159.0 | 168 (11.47)
Weight [Mean (Standard Deviation); unit: kg] | 70.0 (9.19) | 66.2 (11.14) | 71.7 (18.32) | 79.7 (18.30) | 77.6 (18.55) | 70.2 (19.12) | 72.3 (24.39) | 82.3 (24.18) | 87.3 (18.24) | 77.6 (23.65) | 88.4 (36.32) | 84.8 (5.85) | 66.3 (19.90) | 58.0 | 75.69 (19.82)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is a measure of body fat based on height and weight that applies to adult men and women.
  kg/m^2 | 25.2 (4.34) | 22.3 (3.68) | 24.8 (5.00) | 29.5 (6.83) | 26.1 (4.62) | 25.5 (3.51) | 24.3 (5.10) | 26.6 (3.12) | 28.8 (4.85) | 26.7 (7.73) | 27.2 (10.69) | 30.6 (3.27) | 25.5 (6.46) | 22.9 | 26.36 (5.75)
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG performance status measured on 6 point scale to assess participant's performance status. 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=Ambulatory (greater than [>]50% of waking hours), capable of all self care, unable to carry out any work activities
  Participants
    ECOG - 0 | 0 | 2 | 3 | 1 | 0 | 2 | 1 | 0 | 5 | 1 | 2 | 1 | 3 | 1 | 22
    ECOG - 1 | 4 | 3 | 3 | 4 | 3 | 2 | 3 | 3 | 3 | 7 | 2 | 3 | 7 | 0 | 47
    ECOG - >=2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Treatment-emergent Adverse Event (TEAE)
Description: TEAE is defined as an adverse event reported for the first time or worsening of a pre-existing event after the first dose of study treatment.
Time Frame: up to 30 days
Population: The safety population included all enrolled participants who received at least 1 dose of INCB054329.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 / Treatment Group A: 15 MG QD INCB054329 | Part 1 / Treatment Group A: 22.5 MG QD INCB054329 | Part 1 / Treatment Group A: 15 MG BID INCB054329 | Part 1 / Treatment Group A: 30 MG QD INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 5/2 INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 4/3 INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 7/7 INCB054329 | Part 1 / Treatment Group A: 20 MG BID INCB054329 | Part 1 / Treatment Group A: 25 MG BID 5/2 INCB054329 | Part 1 / Treatment Group A: 25 MG BID 7/7 INCB054329 | Part 1 / Treatment Group B: 20 MG BID INCB054329 | Part 2 / Treatment Group A: 20 MG BID INCB054329 | Part 2 / Treatment Group C: 20 mg BID INCB054329
Number analyzed (Participants) | 4 | 5 | 6 | 5 | 3 | 4 | 4 | 3 | 8 | 8 | 4 | 4 | 10 | 1
Participants | 4 | 5 | 6 | 5 | 3 | 4 | 4 | 3 | 8 | 8 | 3 | 4 | 10 | 1

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) Analysis of INCB054329
Description: Cmax is defined as the maximum observed serum concentration measured at steady state (Day 15).
  Study drug was administered with 240 mL of water. Summary of Steady-State, Day 15, was evaluated by dosing regimen.
Time Frame: Summary of steady-state PK parameters by dosing regimen at Day 15
Population: All enrolled patients who received at least 1 dose of study medication and provided at least 1 plasma sample were included.
Measure: Mean (Standard Deviation); unit: nM
Groups:
- INCB054329 Monotherapy - 15 mg QD; INCB054329 Monotherapy - 15 mg BID; INCB054329 Monotherapy - 22.5 mg QD; INCB054329 Monotherapy - 30 mg QD; INCB054329 Monotherapy - 20 mg BID; INCB054329 Monotherapy - 22.5 mg BID; INCB054329 Monotherapy - 25 mg BID; INCB054329 Monotherapy - Overall Dosing Regimen: INCB054329 Monotherapy
Arm/Group | INCB054329 Monotherapy - 15 mg QD | INCB054329 Monotherapy - 15 mg BID | INCB054329 Monotherapy - 22.5 mg QD | INCB054329 Monotherapy - 30 mg QD | INCB054329 Monotherapy - 20 mg BID | INCB054329 Monotherapy - 22.5 mg BID | INCB054329 Monotherapy - 25 mg BID | INCB054329 Monotherapy - Overall Dosing Regimen
Number analyzed (Participants) | 4 | 5 | 4 | 4 | 14 | 12 | 8 | 51
nM | 278 (82.6) | 267 (201) | 479 (154) | 389 (393) | 652 (348) | 720 (472) | 449 (335) | NA (NA) — Dose dependent parameter and overall summary not provided.

3. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) Analysis of INCB054329
Description: Tmax is the time to maximum (peak) drug serum concentration. Study drug was administered with 240 mL of water. Summary of Steady-State, Day 15, was evaluated by dosing regimen.
Time Frame: Summary of steady-state PK parameters by dosing regimen at Day 15
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | INCB054329 Monotherapy - 15 mg QD | INCB054329 Monotherapy - 15 mg BID | INCB054329 Monotherapy - 22.5 mg QD | INCB054329 Monotherapy - 30 mg QD | INCB054329 Monotherapy - 20 mg BID | INCB054329 Monotherapy - 22.5 mg BID | INCB054329 Monotherapy - 25 mg BID | INCB054329 Monotherapy - Overall Dosing Regimen
Number analyzed (Participants) | 4 | 5 | 4 | 4 | 14 | 12 | 8 | 51
hour | 1.0 [0.52 to 1.0] | 0.93 [0.5 to 1.1] | 0.53 [0.5 to 1.0] | 1.0 [0.52 to 1.0] | 1.0 [0.48 to 2.0] | 1.0 [0.5 to 4.1] | 0.77 [0.50 to 2.2] | 1.0 [0.48 to 4.1]

4. Secondary Outcome: Minimum Observed Plasma Concentration Over the Dose Interval (Cmin) Analysis of INCB054329
Description: Minimum observed plasma concentration measured at steady state (Day 15). Study drug was administered with 240 mL of water. Summary of Steady-State, Day 15, was evaluated by dosing regimen.
Time Frame: Summary of steady-state PK parameters by dosing regimen at Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | INCB054329 Monotherapy - 15 mg QD | INCB054329 Monotherapy - 15 mg BID | INCB054329 Monotherapy - 22.5 mg QD | INCB054329 Monotherapy - 30 mg QD | INCB054329 Monotherapy - 20 mg BID | INCB054329 Monotherapy - 22.5 mg BID | INCB054329 Monotherapy - 25 mg BID | INCB054329 Monotherapy - Overall Dosing Regimen
Number analyzed (Participants) | 4 | 5 | 4 | 4 | 13 | 12 | 7 | 49
nM | 0.538 (1.08) | 1.09 (2.45) | 0 (0) | 1.51 (3.02) | 54.2 (91.1) | 14.6 (45) | 0 (0) | NA (NA) — Dose dependent parameter and overall summary not provided.

5. Secondary Outcome: AUC0-t Analysis of INCB054329
Description: AUC0-t is the area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t measured at steady state (Day 15).
  Study drug was administered with 240 mL of water.
Time Frame: Summary of steady-state PK parameters by dosing regimen at Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nM*h
Arm/Group | INCB054329 Monotherapy - 15 mg QD | INCB054329 Monotherapy - 15 mg BID | INCB054329 Monotherapy - 22.5 mg QD | INCB054329 Monotherapy - 30 mg QD | INCB054329 Monotherapy - 20 mg BID | INCB054329 Monotherapy - 22.5 mg BID | INCB054329 Monotherapy - 25 mg BID | INCB054329 Monotherapy - Overall Dosing Regimen
Number analyzed (Participants) | 4 | 5 | 4 | 4 | 14 | 12 | 8 | 51
nM*h | 686 (178) | 611 (628) | 883 (409) | 1150 (1660) | 2130 (1690) | 1970 (1560) | 995 (843) | NA (NA) — Dose dependent parameter and overall summary not provided.

6. Secondary Outcome: Cl/F Analysis of INCB054329
Description: Cl/F is the apparent oral dose clearance measured at steady state (Day 15). Study drug was administered with 240 mL of water.
Time Frame: Summary of steady-state PK parameters by dosing regimen at Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | INCB054329 Monotherapy - 15 mg QD | INCB054329 Monotherapy - 15 mg BID | INCB054329 Monotherapy - 22.5 mg BID | INCB054329 Monotherapy - 30 mg QD | INCB054329 Monotherapy - 20 mg BID | INCB054329 Monotherapy - 22.5 mg QD | INCB054329 Monotherapy - 25 mg BID | INCB054329 Monotherapy - Overall Dosing Regimen
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 14 | 11 | 7 | 48
L/h | 61.8 (21.3) | 85.0 (42.9) | 81.7 (29.4) | 234 (184) | 92.3 (201) | 48.3 (33.7) | 130 (127) | 95.5 (135)

7. Secondary Outcome: Pharmacodynamics (PD) Analysis - Total c-Myc % Inhibition Versus INCB054329
Description: The half maximal inhibitory concentration (IC50) of INCB054329 was measured. The maximal inhibition of total c-Myc was correlated to the level of drug exposure and demonstrated a high degree of interparticipant variability, parallel to the PK data.
  The measure was performed as a value across all cohorts. The entire dose escalation data set was used to create the relationship curve. Analysis of individual cohorts contained too few subjects and was biased toward one region of the curve so that the relationship was poorly defined.
  Individual data points from all subjects were subjected to a nonlinear least squares regression analysis with no weighting, resulting in a sigmoidal dose response curve defining the relationship. The numerical value given is the projected INCB0054329 concentration in nM that produced 50% inhibition of c-myc expression.
Time Frame: Day 15 in all cohorts
Population: Individual data points from all subjects were subjected to a nonlinear least squares regression analysis with no weighting, resulting in a sigmoidal dose response curve defining the relationship. The numerical value given is the projected INCB0054329 concentration in nM that produced 50% inhibition of c-myc expression.
Measure: Number; unit: nM
Arm/Group | INCB054329 Monotherapy
Number analyzed (Participants) | 49
nM | 283.4

8. Secondary Outcome: Objective Response Rate (ORR)
Description: Defined as the percentage of subjects having complete response (CR) or partial response (PR). The best overall response was defined as the best response recorded before and including the first event of Progressive disease (PD).
Time Frame: Baseline through end of study, up to 6 months
Population: As a result of early termination of the study, only participants in Part 2 of the study were evaluated; Treatment Group C was not evaluated due to early termination from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 / Treatment Group A: 20 MG BID INCB054329 | Part 2 / Treatment Group C: 20 mg BID INCB054329
Number analyzed (Participants) | 10 | 0
Participants
  Complete response (CR) | 0 |
  Partial response (PR) | 0 |
  Stable disease (SD) >= 6 months | 0 |
  Stable disease (SD) < 6 months | 4 |
  Progressive disease (PD) | 5 |
  Not evaluable (NE) | 1 |

9. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time from earliest date of disease response until earliest date of disease progression or death.
Time Frame: Baseline through end of study, up to 6 months
Population: As a result of early termination of the study, there are no participants that are responders and therefore DOR was not achieved.
Arm/Group | Part 1 / Treatment Group A: 15 MG QD INCB054329 | Part 1 / Treatment Group A: 22.5 MG QD INCB054329 | Part 1 / Treatment Group A: 15 MG BID INCB054329 | Part 1 / Treatment Group A: 30 MG QD INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 5/2 INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 4/3 INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 7/7 INCB054329 | Part 1 / Treatment Group A: 20 MG BID INCB054329 | Part 1 / Treatment Group A: 25 MG BID 5/2 INCB054329 | Part 1 / Treatment Group A: 25 MG BID 7/7 INCB054329 | Part 1 / Treatment Group B: 20 MG BID INCB054329 | Part 2 / Treatment Group A: 20 MG BID INCB054329 | Part 2 / Treatment Group C: 20 mg BID INCB054329
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is the time from start of study treatment to first documentation of progression, or to death due to any cause, whichever comes first
Time Frame: Baseline through end of study, up to 6 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2 / Treatment Group A: 20 MG BID INCB054329 | Part 2 / Treatment Group C: 20 mg BID INCB054329
Number analyzed (Participants) | 10 | 0
months | 2.04 [0.63 to 4.21] |

11. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of the participant's death.
Time Frame: Baseline through end of study, up to 6 months for participants in Part 2
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2 / Treatment Group A: 20 MG BID INCB054329 | Part 2 / Treatment Group C: 20 mg BID INCB054329
Number analyzed (Participants) | 10 | 0
months | 7.09 [3.13 to NA] — The upper CI limit of median PFS could not be estimated by the Brookmeyer and Crowley method because there were not enough events. |

ADVERSE EVENTS:
Time Frame: From the first dose of study medication up to 6 months or up to study termination date 31Jan2018. Follow-up data included up until database lock 11APR2018.
Description: The safety evaluable population consisted of all participants exposed to at least 1 dose of study drug.
Arm/Group | Part 1 / Treatment Group A: 15 MG QD INCB054329 | Part 1 / Treatment Group A: 22.5 MG QD INCB054329 | Part 1 / Treatment Group A: 15 MG BID INCB054329 | Part 1 / Treatment Group A: 30 MG QD INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 5/2 INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 4/3 INCB054329 | Part 1 / Treatment Group A: 22.5 MG BID 7/7 INCB054329 | Part 1 / Treatment Group A: 20 MG BID INCB054329 | Part 1 / Treatment Group A: 25 MG BID 5/2 INCB054329 | Part 1 / Treatment Group A: 25 MG BID 7/7 INCB054329 | Part 1 / Treatment Group B: 20 MG BID INCB054329 | Part 2 / Treatment Group A: 20 MG BID INCB054329 | Part 2 / Treatment Group C: 20 mg BID INCB054329
All-Cause Mortality (participants affected / at risk) | 4/4 | 4/5 | 3/6 | 4/5 | 2/3 | 2/4 | 3/4 | 1/3 | 6/8 | 6/8 | 3/4 | 2/4 | 6/10 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/5 | 1/6 | 1/5 | 3/3 | 3/4 | 1/4 | 1/3 | 3/8 | 3/8 | 1/4 | 3/4 | 3/10 | 1/1
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 6/6 | 5/5 | 3/3 | 4/4 | 4/4 | 3/3 | 8/8 | 8/8 | 2/4 | 4/4 | 10/10 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 / Treatment Group A: 15 MG QD INCB054329 (N=4) | Part 1 / Treatment Group A: 22.5 MG QD INCB054329 (N=5) | Part 1 / Treatment Group A: 15 MG BID INCB054329 (N=6) | Part 1 / Treatment Group A: 30 MG QD INCB054329 (N=5) | Part 1 / Treatment Group A: 22.5 MG BID INCB054329 (N=3) | Part 1 / Treatment Group A: 22.5 MG BID 5/2 INCB054329 (N=4) | Part 1 / Treatment Group A: 22.5 MG BID 4/3 INCB054329 (N=4) | Part 1 / Treatment Group A: 22.5 MG BID 7/7 INCB054329 (N=3) | Part 1 / Treatment Group A: 20 MG BID INCB054329 (N=8) | Part 1 / Treatment Group A: 25 MG BID 5/2 INCB054329 (N=8) | Part 1 / Treatment Group A: 25 MG BID 7/7 INCB054329 (N=4) | Part 1 / Treatment Group B: 20 MG BID INCB054329 (N=4) | Part 2 / Treatment Group A: 20 MG BID INCB054329 (N=10) | Part 2 / Treatment Group C: 20 mg BID INCB054329 (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 / Treatment Group A: 15 MG QD INCB054329 (N=4) | Part 1 / Treatment Group A: 22.5 MG QD INCB054329 (N=5) | Part 1 / Treatment Group A: 15 MG BID INCB054329 (N=6) | Part 1 / Treatment Group A: 30 MG QD INCB054329 (N=5) | Part 1 / Treatment Group A: 22.5 MG BID INCB054329 (N=3) | Part 1 / Treatment Group A: 22.5 MG BID 5/2 INCB054329 (N=4) | Part 1 / Treatment Group A: 22.5 MG BID 4/3 INCB054329 (N=4) | Part 1 / Treatment Group A: 22.5 MG BID 7/7 INCB054329 (N=3) | Part 1 / Treatment Group A: 20 MG BID INCB054329 (N=8) | Part 1 / Treatment Group A: 25 MG BID 5/2 INCB054329 (N=8) | Part 1 / Treatment Group A: 25 MG BID 7/7 INCB054329 (N=4) | Part 1 / Treatment Group B: 20 MG BID INCB054329 (N=4) | Part 2 / Treatment Group A: 20 MG BID INCB054329 (N=10) | Part 2 / Treatment Group C: 20 mg BID INCB054329 (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 3 | 3 | 1 | 0 | 2 | 3 | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 2 | 1 | 2 | 0 | 3 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 2 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 1 | 2 | 1 | 2 | 5 | 5 | 1 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 2 | 4 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 3 | 1 | 3 | 2 | 3 | 2 | 2 | 4 | 1 | 1 | 2 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 2 | 1 | 2 | 1 | 0
Pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 3 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 3 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 0 | 1 | 1 | 1 | 3 | 1 | 3 | 0 | 1 | 3 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 1 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 2 | 0 | 1 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT02431260/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT02431260/SAP_001.pdf